CLINICAL TRIAL: NCT04744090
Title: The Potential Anti-inflammatory Effect of Roflumilast as Add-on Therapy in The Management of Hospitalized Patients With Mild Acute Respiratory Distress Syndrome
Brief Title: Roflumilast as add-on Therapy in Early Cases of ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Abdel Moniem Abdel Rasheed, Professor Emeritus, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-292-2020
Record Dates: First submitted 2021-01-16; First posted 2021-02-08 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast add-on (Experimental): Eligible patients will take 500 Mcg of roflumilast once daily (up to 28 days) plus standard of care.
  Interventions: Drug: Roflumilast
- Placebo control (Placebo Comparator): Eligible patients will take placebo plus standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 1. Roflumilast 500 mcg daily for up to 28 days
  2. Total follow up time will be 28 days.
  3. Proinflammatory parameters will be assessed at baseline, day 7, day 14, and at the end of treatment.
  4. Roflumilast will be combined with standard of care for ARDS.
  5. During hospitalization, clinical and laboratory data will be recorded daily in the medical history of the patient and in data collection table of the study.
  6. During hospitalization, adverse drug reaction will be monitored clinically and by laboratory tests.
  7. In case of an adverse effect or a need to discontinue the treatment, roflumilast should be suspended.
  Arms: Roflumilast add-on
Drug: Placebo — Placebo (identical to roflumilast dosage form) will be used for placebo-comparator group.
  Arms: Placebo control

SUMMARY:
* Mild cases of ARDS will be included in a two-arm protocol, to receive 500 mcg of roflumilast daily up to 28 days (FDA approved dose for COPD) plus standard of care versus standard of care alone.
* Approximately 76 hospitalized patients with ARDS will be enrolled in this study.
* Eligible patients will be randomized at ratio of (1:1) to receive either roflumilast plus standard of care or standard of care alone.

DETAILED DESCRIPTION:
• Methodology in details:

* Informed consent will be obtained from included participants.
* Mild cases of ARDS will be included in a two-arm protocol, to receive 500 mcg of roflumilast daily up to 28 days (FDA approved dose for COPD) plus standard of care versus standard of care alone.
* Approximately 76 hospitalized patients with ARDS will be enrolled in this study.
* Eligible patients will be randomized at ratio of (1:1) to receive either roflumilast plus standard of care or standard of care alone.
* Randomization:

Randomization will be in 1:1 ratio using permuted blocks of different sizes. Random.org website will be used for random selection of a sequence of blocks. The latter will be used to generate a randomized list which will be generated and stored by a third party independent of the study team. For allocation concealment, the list will be used to make sequentially numbered sealed opaque envelopes, each containing the sequential randomization number and allocation of subsequent cases. Envelopes will be handed to the study team member responsible for medication preparation. Each envelope will be opened only after:

1. Screening for eligibility
2. Obtaining consent
3. Recording baseline characters The treatment allocation dictated in the envelope will be documented in the case record form and will be subject to audit to assure correct randomization according to the original list.

   * Intervention:

Drug: Roflumilast

1. Roflumilast 500 mcg daily for up to 28 days
2. Total follow up time will be 28 days.
3. Proinflammatory parameters will be assessed at baseline, day 7, day 14, and at the end of treatment.
4. Roflumilast will be combined with standard of care for ARDS.
5. During hospitalization, clinical and laboratory data will be recorded daily in the medical history of the patient and in data collection table of the study.
6. During hospitalization, adverse drug reaction will be monitored clinically and by laboratory tests.
7. In case of an adverse effect or a need to discontinue the treatment, roflumilast should be suspended.

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign informed consent
* Patients >18 years old male or female
* Mild cases of ARDS according to the Berlin criteria (PaO/FiO 200 to 300 mmHg)

Exclusion Criteria:

* Pregnancy and breast feeding
* History of hypersensitivity to roflumilast
* Patients with mechanical respiratory assistance (severe ARDS)
* Patients under treatment with roflumilast for COPD
* Patients with psychiatric diseases
* Hepatic cirrhosis (Child-Pugh score B or C)
* Refused to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in clinical picture (two-point reduction in patient's admission status) | Follow up for up to 28 days.
  Defined as a two-point reduction in patient's admission status on a five-point ordinal scale, or live discharge from hospital whichever came first.
  • The five-point ordinal scale is as follow:
  1. Discharge
  2. Hospital admission, not requiring oxygen supplement
  3. Hospital admission, requiring oxygen supplement
  4. Hospital admission for high flow oxygen therapy or non-invasive mechanical ventilation
  5. Hospital admission for mechanical ventilation or extracorporeal membrane oxygenation

SECONDARY OUTCOMES:
Evaluation of change in systemic inflammatory parameters, including ferritin. | Weekly assessment (baseline, day7, day14, at the end) for up to 28 days.
Evaluation of change in systemic inflammatory parameters, including CRP. | Weekly assessment (baseline, day7, day14, at the end) for up to 28 days.
Evaluation of change in systemic inflammatory parameters, including LDH. | Weekly assessment (baseline, day7, day14, at the end) for up to 28 days.
Total hospital stay. | Follow up for up to 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Abdel Rasheed, Professor, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Misr International Hospital, Giza, Doki
  - Cairo University Hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No